CLINICAL TRIAL: NCT04452721
Title: Prognosis Factors for the Treatment of Pectus Carinatum With a Dynamic Compression System
Acronym: Pectusdyn
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH030
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pectus Carinatum
Keywords: Pectus Carinatum; Dynamic compression system
MeSH Terms: conditions — Pectus Carinatum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: 340 to 400 patients
  Interventions: Other: dynamic compression system
- Validation cohort: 120 patients
  Interventions: Other: dynamic compression system

INTERVENTIONS:
Other: dynamic compression system — It is a harness that the patient wears all day long for an average duration of 1 year, and that remodels the chest by exerting a moderate pressure on it

SUMMARY:
Pectus carinatum is a deformation of the thoracic wall causing an aesthetic prejudice. Since 2011, our team uses a dynamic compression system to treat this deformation. It is a harness that the patient wears all day long for an average duration of 1 year, and that remodels the chest by exerting a moderate pressure on it. The local cohort is one of the largest in the world. The few previous publications have shown the validity of this method, but the prognosis factors for success of this innovative treatment are not yet identified.

DETAILED DESCRIPTION:
The principal insvestigator hypothesizes that the success or failure of the treatment depends on several parameters assessable before treatment, such as the patient's age, gender, initial correction pressure, symmetry or not of the deformation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received proper information about the study.
* Patient with clinically diagnosed pectus carinatum.
* Treated at Saint-Etienne University Hospital using a dynamic compression system.
* Between October 2011 and January 2020 for the retrospective part, then between January 2020 and January 2022 for the validation cohort.
* With more than 6 months of follow-up since the beginning of the treatment.

Exclusion Criteria:

-

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Refusal to participate to this treatment
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Decrease of the deformation of more than 50% (measured in mm) after 6 months of treatment | After 6 months of treatment
  Dynamic compression system

SECONDARY OUTCOMES:
Failure of treatment assessed by the patient, ie if the patients considers the treatment to have failed, if he choose to underwent surgery afterwards, or if he considered the pectus carinatum to have relapsed | After the end of treatment (6 months to 2 years)
  Dynamic compression system

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien SCALABRE, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kieffer De Marco L, Filaire L, Vermersch S, Chapelle C, Garcin A, Tiffet O, Scalabre A. Prognostic Factors for Pectus Carinatum Treated by Dynamic Compression System: PECTUSDYN Trial. Eur J Cardiothorac Surg. 2026 Jan 6;68(1):ezaf444. doi: 10.1093/ejcts/ezaf444. PMID 41390917